

## **Statistical Analysis Plan**

**BI Trial No.:** 0352-2119

Title: Digital Auscultation Test - Development of an Innovative

Approach - using modern technologies - to improve the diagnosis

of rare lung diseases – expanded data collection Idiopathic

Pulmonary Fibrosis.

Investigational

product(s):

Not applicable

Responsible trial statistician:

Tel:

Fax:

Date of statistical

analysis plan:

26 JUL 2018

Version: Final

Page 1 of 9

### **Proprietary confidential information**

© 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

TSAP for BI Trial No: 0352.2119

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## TABLE OF CONTENTS

| TITI | E PA | GE | 1 |
|------------|--------|-------------------------------------------------|---|
| 1. | TA] | GEBLE OF CONTENTS | 2 |
| | | ABLES | |
| 2. | | T OF ABBREVIATIONS | |
| <b>3.</b> | | TRODUCTION | |
| <b>4.</b> | | ANGES IN THE PLANNED ANALYSIS OF THE STUDY | |
| 5. | | TCOMES | |
| s.<br>5.1 | | RIMARY OUTCOMES | |
| 5.1<br>5.2 | | ECONDARY OUTCOMES | |
| 5.3 | | THER OUTCOMES. | |
| 6. | | NERAL ANALYSIS DEFINITIONS | |
| o.<br>6.1 | | XPOSURE | |
| 6.2 | I | MPORTANT PROTOCOL VIOLATIONS | 4 |
| 6.3 | | ATIENT SETS ANALYSED | |
| | 6.3.1 | All Subjects Enrolled Set (ENR) | |
| 6.5 | | OOLING OF CENTRES | |
| 6.6 | | ANDLING OF MISSING DATA AND OUTLIERS | |
| <b>6.7</b> | | ASELINE, TIME WINDOWS AND CALCULATED VISITS | |
| <b>7.</b> | | ANNED ANALYSIS | |
| <b>7.1</b> | | EMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | |
| 7.2 | | ONCOMITANT DISEASES AND MEDICATION | |
| 7.3 | | REATMENT ADHERENCE | |
| 7.4 | | IETHODS ADDRESSING BIAS | 6 |
| 7.5 | | IETHODS ADDRESSING CONFOUNDING / EFFECT MEASURE | |
| 7.6 | | IODIFICATIONRIMARY ANALYSES | |
| 7.6<br>7.7 | | ECONDARY ANALYSES | |
| 7.7<br>7.8 | | THER ANALYSES. | |
| 7.9 | _ | XPOSURE TIME | |
| 7.1 | | AFETY ANALYSIS. | |
| | 7.10.1 | Adverse events | |
| , | 7.10.2 | Laboratory data | |
| , | 7.10.3 | Vital signs | 7 |
| , | 7.10.4 | ECG | 7 |
| | 7.10.5 | Others | |
| <b>7.1</b> | | NTERIM ANALYSES | |
| 8. | RE | FERENCES | 7 |
| 10 | HIS | STORY TABLE | 9 |

#### LIST OF TABLES

Not applicable.

## 1. LIST OF ABBREVIATIONS

| AE | Adverse Event |
|--------|------------------------------------------------|
| BI | Boehringer Ingelheim |
| BMI | Body Mass Index |
| CRF | Case Report Form |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CTP | Clinical Trial Protocol |
| ECG | Electrocardiography |
| EMA | European Medicines Agency |
| ENMST | All Subjects Entered Main-Study Set |
| ENR | All Subjects Enrolled Set |
| ENSST | All Subjects Entered Sub-Study Set |
| ENT | All Subject Entered Set |
| IPF | Idiopathic Pulmonary Fibrosis |
| IRB | Institutional Review Board |
| MedDRA | Medical Dictionary for Regulatory Activities |
| SAE | Serious Adverse Event |
| SOC | System Organ Class |
| SOP | Standard Operating Procedure |
| TCM | Trial Clinical Manager |
| TSAP | Trial Statistical Analysis Plan |

## 2. INTRODUCTION

This TSAP assumes familiarity with the Clinical Trial Protocol (CTP), including Protocol Amendments.

There is no investigational drug being used in this study. Focus will be on two complimentary groups, the one group includes only patients diagnosed with IPF (IPF group) and the other group only includes patients not diagnosed with IPF (non-IPF group).

In addition a sub-study is planned to collect sound recordings using two different electronic stethoscope sequentially from approximately 50 additional patients (approximately 20 patients diagnosed with IPF and approximately 30 diagnosed with a non-IPF lung disease).

SAS® Version xx will be used for all analyses.

TSAP for BI Trial No: 0352.2119

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 3. CHANGES IN THE PLANNED ANALYSIS OF THE STUDY

Not applicable

## 4. OUTCOMES

#### 4.1 PRIMARY OUTCOMES

For each patient the auscultation sound files will be collected at 12 points of the body. The primary outcome will be the percentage collected auscultation point.

## 4.2 SECONDARY OUTCOMES

The secondary outcomes are:

- Patient reported symptoms (8 questions)
- Smoking status
- BMI
- Gender

#### 4.3 OTHER OUTCOMES

The other outcomes are:

- Age
- Height
- Weight
- Blood pressure
- Pulse rate
- Weight loss

## 5. GENERAL ANALYSIS DEFINITIONS

## 5.1 EXPOSURE

Not applicable.

## 5.2 IMPORTANT PROTOCOL VIOLATIONS

For this trial no important protocol violations are defined. However all protocol violations will be listed and tabulated.

TSAP for BI Trial No: 0352.2119 Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### PATIENT SETS ANALYSED

As this is a one visit trial without any trial medication only one patient set will be defined.

#### 5.3.1 All subject enrolled Set (ENR)

The all subject enrolled set will contain all subjects that signed informed consent.

### 5.3.2 All Subjects Entered Set (ENT)

The all subjects entered set will contain all subjects for which visit data is available.

## 5.3.3 All Subjects Entered Main-Study Set (ENMST)

The all subjects entered main study set will contain all subjects for which visit data is available and are not part of the Sub-Study.

#### 5.3.4 All Subjects Entered Sub-Study Set (ENSST)

The all subjects entered sub-study set will contain all subjects for which visit data is available and are part of the Sub-Study.

#### 5.5 **POOLING OF CENTRES**

Not applicable.

#### HANDLING OF MISSING DATA AND OUTLIERS

No imputation for missing data nor for outliers is planned in this trial. Missing or incomplete AE dates will be handled as described in "Handling of missing and incomplete AE dates [1].

## BASELINE, TIME WINDOWS AND CALCULATED VISITS

Not applicable.

#### 6. PLANNED ANALYSIS

All tables will be presented by diagnose group (IPF group and non-IPF group) and overall. At least the following descriptive statistics will be calculated for all continuous endpoints: N, arithmetic mean, standard deviation, minimum, median, maximum.

#### **DISPOSITION**

Only descriptive statistics are planned for this section of the report and will be presented for the ENT set.

#### DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS 6.2

Only descriptive statistics are planned for this section of the report and will be presented for the ENT, ENMST and ENSST set.

#### 6.3 CONCOMITANT DISEASES AND SURGIRICAL PROCEDURES

Only descriptive statistics are planned for this section of the report and will be presented for the ENT, ENMST and ENSST set.

#### 6.4 TREATMENT ADHERENCE

Not applicable.

#### 6.5 METHODS ADDRESSING BIAS

Not applicable.

# 6.6 METHODS ADDRESSING CONFOUNDING / EFFECT MEASURE MODIFICATION

Not applicable

### 6.7 PRIMARY ANALYSES

Only descriptive statistics are planned for this section of the report and will be presented for the ENT, ENMST and ENSST set.

#### 6.8 SECONDARY ANALYSES

Only descriptive statistics are planned for this section of the report and will be presented for the ENT, ENMST and ENSST set.

#### 6.9 OTHER ANALYSES

Only descriptive statistics are planned for this section of the report and will be presented for the ENT, ENMST and ENSST set.

## 6.10 EXPOSURE TIME

Not applicable.

#### 6.11 SAFETY ANALYSIS

All safety analyses will be performed on the ENR set.

#### **6.11.1** Adverse events

Unless otherwise specified, the analyses of adverse events will be descriptive in nature. All analyses of AEs will be based on the number of subjects with AEs and NOT on the number of AEs.

Adverse Events (AEs) will be coded using MedDRA central coding dictionary, Version 21.0 or higher. The system organ classes will be sorted by internationally agreed EMA SOC order (refer to Section 8); preferred terms will be sorted by decreasing frequencies (within system organ class).

For analysis multiple AE occurrence data on the CRF will be collapsed into an AE provided that all of the following applies:

• All AE attributes are identical.

TSAP for BI Trial No: 0352.2119

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

• The occurrences were time-overlapping or time-adjacent (time-adjacency of 2 occurrences is given if the second occurrence started on the same day or on the day after the end of the first occurrence.

For further details on summarization of AE data, please refer to (1, 2).

An overall summary of adverse events will be presented.

The frequency of subjects with adverse events will be summarised by treatment, primary system organ class and preferred term (mention MedDRA levels to be displayed in the tables). Separate tables will be provided for subjects with serious adverse events.

In addition the system organ classes will be sorted alphabetically, preferred terms will be sorted by frequency (within system organ class).

## 6.11.2 Laboratory data

Not applicable.

#### 6.11.3 Vital signs

Only descriptive statistics are planned for this section of the report.

#### 6.11.4 ECG

Not applicable.

#### **6.11.5** Others

Only descriptive statistics are planned for this section of the report.

#### 6.12 INTERIM ANALYSES

Not applicable.

#### 7. REFERENCES

- 1. 001-MCG-156\_RD-01: "Handling of missing and incomplete AE dates", current version; IDEA for CON.
- 2. 001-MCG-156: "Handling and summarization of adverse event data for clinical trial reports and integrated summaries", current version; IDEA for CON.

# 8. EMA SOC ORDER FOR PRESENTATION OF THE AE IN THE TABLES

Order System Organ Class

- 0 Uncoded
- 1 Infections and infestations
- 2 Neoplasms benign, malignant and unspecified (incl cysts and polyps)

- 3 Blood and lymphatic system disorders
- 4 Immune system disorders
- 5 Endocrine disorders
- 6 Metabolism and nutrition disorders
- 7 Psychiatric disorders
- 8 Nervous system disorders
- 9 Eye disorders
- 10 Ear and labyrinth disorders
- 11 Cardiac disorders
- 12 Vascular disorders
- 13 Respiratory, thoracic and mediastinal disorders
- 14 Gastrointestinal disorders
- 15 Hepatobiliary disorders
- 16 Skin and subcutaneous tissue disorders
- 17 Musculoskeletal and connective tissue disorders
- 18 Renal and urinary disorders
- 19 Pregnancy, puerperium and perinatal conditions
- 20 Reproductive system and breast disorders
- 21 Congenital, familial and genetic disorders
- 22 General disorders and administration site conditions
- 23 Investigations
- 24 Injury, poisoning and procedural complications
- 25 Surgical and medical procedures
- 26 Social circumstances
- 27 Product issues

## 9. HISTORY TABLE

Shared; dependent on section changed



#### APPROVAL / SIGNATURE PAGE

Document Number: c24453484 Technical Version Number: 1.0

**Document Name:** 8-01-tsap-core

**Title:** Digital Auscultation Test - Development of an Innovative Approach - using modern technologies - to improve the diagnosis of rare lung diseases – expanded data collection Idiopathic Pulmonary Fibrosis

## **Signatures (obtained electronically)**

| Meaning of Signature | Signed by | <b>Date Signed</b> |
|---------------------------------|-----------|------------------------|
| Author-Trial Statistician | | 26 Jul 2018 15:16 CEST |
| Approval-Trial Clinical Monitor | | 26 Jul 2018 15:22 CEST |
| Approval-Biostatistics | | 27 Jul 2018 01:19 CEST |

Boehringer IngelheimPage 2 of 2Document Number: c24453484Technical Version Number: 1.0

## (Continued) Signatures (obtained electronically)

| Meaning of Signature Signed by Date Signed |
|--------------------------------------------|
|--------------------------------------------|